CLINICAL TRIAL: NCT00003418
Title: Randomized Double-Blind Trial in Postmenopausal Women With Primary Breast Cancer Who Have Received Adjuvant Tamoxifen for 2-3 Years, Comparing Subsequent Adjuvant Exemestane Treatment With Further Tamoxifen
Brief Title: Exemestane Compared With Tamoxifen in Treating Postmenopausal Women With Primary Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Collaborative Cancer Group (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); UNICANCER (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066434; ICCG-96OEXE031-C1396-BIG9702; EORTC-10967; FRE-FNCLCC-PACS02/96OEXE031; EU-20013; EU-99002; ICCG-BIG-97/02
Record Dates: First submitted 1999-11-01; First posted 2004-01-23 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2008-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage III breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Tamoxifen

INTERVENTIONS:
Drug: exemestane
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using exemestane or tamoxifen may fight breast cancer by blocking the uptake of estrogen. It is not yet known whether exemestane is more effective than tamoxifen in treating breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of exemestane with that of tamoxifen in treating postmenopausal women with primary breast cancer who have already received 2-3 years of tamoxifen following surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare, in terms of disease-free survival and overall survival, the sequential administration of exemestane with administration of further tamoxifen until 5 years of therapy is achieved in postmenopausal women with operable breast cancer who have already received 2-3 years of adjuvant tamoxifen. II. Compare the regimens in terms of the incidence of contralateral breast cancer and long term tolerability of the regimens in these patients. III. Determine the tolerability of each regimen in terms of endometrial status, bone metabolism, lipid profile, and coagulation profile in these patients. IV. Assess quality of life in these patients treated with these regimens.

OUTLINE: This is a randomized, double blind, multicenter study. Following 2-3 years of adjuvant treatment with tamoxifen, patients are randomized to receive either oral tamoxifen daily or oral exemestane daily for the remainder of the 5 year period in the absence of disease relapse or unacceptable toxicity. Quality of life is assessed at some centers. Patients are followed at least every 3 months for the first year of treatment, every 6 months for the next two years and then annually thereafter until year 10.

PROJECTED ACCRUAL: Approximately 4400 patients (2200 patients in each arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: At diagnosis: Histologically confirmed unilateral adenocarcinoma of the breast that was considered operable Must have had adequate therapy for primary disease including chemotherapy/ovarian ablation if appropriate and local postoperative radiotherapy if the patient received conservative (breast preserving) surgery Must have remained disease-free after therapy for primary disease Must have been receiving tamoxifen for minimum of 2 years and maximum of 3 years 1 month with no more than 1 month break at any one time No inflammatory breast cancer, histologically positive supraclavicular nodes, or ulceration/infiltration or skin metastases No evidence of local relapse or distant metastasis (on chest x-ray, scintigraphic bone scanning and liver ultrasonography/CT scanning) at any time Hormone receptor status: Estrogen receptor positive or unknown

PATIENT CHARACTERISTICS: Age: Postmenopausal as defined below Sex: Female Menopausal status: Postmenopausal as defined by: 55 years of age and over, and amenorrhea for greater than 2 years OR Radiation menopause (at least 3 months previously) or surgical oophorectomy OR Natural amenorrhea for at least 1 year at breast cancer diagnosis Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 Hemoglobin normal Hepatic: SGOT no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No significant cardiac disorder Other: No significant skeletal or endocrine disorders No clinical evidence of severe osteoporosis and/or history of osteoporotic fracture No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix No psychiatric or addictive disorders

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Prior or concurrent bisphosphonates allowed Adjuvant or neoadjuvant chemotherapy for primary disease allowed Endocrine therapy: At least 4 weeks since prior hormone replacement therapy (oral, topical, or vaginal) Prior low-dose progestins for relief of menopausal symptoms (up to 6 months duration) allowed No concurrent progestins No concurrent systemic corticosteroids for a prolonged period (i.e., greater than 2 weeks) No concurrent selective estrogen receptor modulators Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics Other: Prior participation and completion of therapy on another clinical study of systemic therapy (e.g., comparison of chemotherapy schedules) allowed No concurrent warfarin Concurrent treatment for other diseases allowed only when clinically indicated

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4400 (Estimated)
Dates: Start 1998-02

CONTACTS AND LOCATIONS:
Overall Officials: R. Charles Coombes, MD, MRCP, FRCP, PhD, FMedSci, Study Chair — Charing Cross Hospital; Robert Paridaens, MD, PhD, Study Chair — University Hospital, Gasthuisberg; Moise Namer, MD, PhD, Study Chair — Centre Antoine Lacassagne
Locations (3):
- U.Z. Gasthuisberg, Leuven, Belgium
- Centre Antoine Lacassagne, Nice, France
- Charing Cross Hospital, London, England, United Kingdom

REFERENCES:
- [Result] Coleman RE, Banks LM, Girgis SI, Kilburn LS, Vrdoljak E, Fox J, Cawthorn SJ, Patel A, Snowdon CF, Hall E, Bliss JM, Coombes RC; Intergroup Exemestane Study group. Skeletal effects of exemestane on bone-mineral density, bone biomarkers, and fracture incidence in postmenopausal women with early breast cancer participating in the Intergroup Exemestane Study (IES): a randomised controlled study. Lancet Oncol. 2007 Feb;8(2):119-27. doi: 10.1016/S1470-2045(07)70003-7. PMID 17267326
- [Result] Coombes RC, Kilburn LS, Snowdon CF, Paridaens R, Coleman RE, Jones SE, Jassem J, Van de Velde CJ, Delozier T, Alvarez I, Del Mastro L, Ortmann O, Diedrich K, Coates AS, Bajetta E, Holmberg SB, Dodwell D, Mickiewicz E, Andersen J, Lonning PE, Cocconi G, Forbes J, Castiglione M, Stuart N, Stewart A, Fallowfield LJ, Bertelli G, Hall E, Bogle RG, Carpentieri M, Colajori E, Subar M, Ireland E, Bliss JM; Intergroup Exemestane Study. Survival and safety of exemestane versus tamoxifen after 2-3 years' tamoxifen treatment (Intergroup Exemestane Study): a randomised controlled trial. Lancet. 2007 Feb 17;369(9561):559-70. doi: 10.1016/S0140-6736(07)60200-1. PMID 17307102
- [Result] Coombes RC, Paridaens R, Jassem J, et al.: First mature analysis of the Intergroup Exemestane Study. [Abstract] J Clin Oncol 24 (Suppl 18): A-LBA527, 2006.
- [Result] Coombes RC, Hall E, Gibson LJ, Paridaens R, Jassem J, Delozier T, Jones SE, Alvarez I, Bertelli G, Ortmann O, Coates AS, Bajetta E, Dodwell D, Coleman RE, Fallowfield LJ, Mickiewicz E, Andersen J, Lonning PE, Cocconi G, Stewart A, Stuart N, Snowdon CF, Carpentieri M, Massimini G, Bliss JM, van de Velde C; Intergroup Exemestane Study. A randomized trial of exemestane after two to three years of tamoxifen therapy in postmenopausal women with primary breast cancer. N Engl J Med. 2004 Mar 11;350(11):1081-92. doi: 10.1056/NEJMoa040331. PMID 15014181